CLINICAL TRIAL: NCT07270094
Title: Effect of Dual Task in Aquatic Physical Therapy in Older Adults: A Randomized Controlled Trial
Brief Title: Effect of Dual Task in Aquatic Physical Therapy in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Leiria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CE/IPLEIRIA/47/2025
Record Dates: First submitted 2025-11-18; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Healthy Older Adults
Keywords: Aquatic physiotherapy; Dual task; Older adults; Cognitive function; Functional mobility; Balance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquatic Dual-Task Training (GDTA) (Experimental): A 12-week aquatic dual-task training program, consisting of two 45-minute sessions per week, combining motor exercises with concurrent cognitive tasks.
  Interventions: Behavioral: Aquatic Dual-Task Training
- Conventional Aquatic Exercise (GEAC) (Active Comparator): A 12-week aquatic exercise program, consisting of two 45-minute sessions per week, including standard therapeutic aquatic exercises without cognitive dual-task components.
  Interventions: Behavioral: Conventional Aquatic Exercise

INTERVENTIONS:
Behavioral: Aquatic Dual-Task Training — Participants perform a structured aquatic exercise program including mobility, balance, and functional strengthening tasks.
  In the experimental arm, each motor task is performed simultaneously with a cognitive task (dual-task condition), including attention, memory, and executive-function challenges (e.g., verbal fluency, counting backwards, category switching).
  Arms: Aquatic Dual-Task Training (GDTA)
Behavioral: Conventional Aquatic Exercise — Participants perform the same structured aquatic exercise program as the experimental group, including mobility, balance, and functional strengthening tasks, but without the addition of cognitive challenges.
  Exercises are performed in a single-task motor condition, representing standard aquatic physiotherapy practice.
  Arms: Conventional Aquatic Exercise (GEAC)

SUMMARY:
Population ageing is associated with declines in motor and cognitive functions, which compromise autonomy and increase the risk of falls and cognitive impairment. Dual-task training programs have demonstrated additional benefits for physical and cognitive health compared with motor exercise alone. Aquatic environments provide unique advantages for older adults, facilitating movement execution and increasing adherence. However, evidence comparing aquatic dual-task training with conventional aquatic exercise remains scarce.

This randomized, controlled, double-blind trial aims to compare the effects of an aquatic dual-task training program with those of a conventional aquatic exercise program on cognitive and motor functions in cognitively preserved older adults. Eighty-four participants aged 65 years or older were recruited, screened for eligibility, and randomly assigned to one of two groups: the Dual-Task Aquatic Group (n = 42) or the Conventional Aquatic Exercise Group (n = 42). The 12-week intervention consisted of two weekly sessions of 45 minutes. Cognitive (Montreal Cognitive Assessment; Mini-Mental State Examination) and motor outcomes (Timed Up and Go Test; Berg Balance Scale) were assessed pre- and post-intervention. Statistical analyses included intra- and inter-group comparisons using non-parametric tests, with a significance level of 5%.

The dual-task group demonstrated significant improvements in balance, functional mobility, and cognitive performance, while the control group showed improvements only in motor outcomes. Between-group comparisons revealed superior cognitive gains in the dual-task group, with no differences in motor outcomes. Adherence exceeded 95% in both groups.

DETAILED DESCRIPTION:
Population ageing introduces challenges associated with progressive motor and cognitive decline, increasing dependence, fall risk, and vulnerability to neurocognitive disorders. Dual-task training-combining simultaneous motor and cognitive tasks-has shown promising benefits in older adults, outperforming isolated motor exercise in several domains. The aquatic environment presents additional therapeutic advantages such as reduced joint load, enhanced balance safety, and increased adherence. Despite these strengths, few studies have rigorously compared aquatic dual-task training with conventional aquatic exercise.

This randomized, controlled, double-blind trial investigates the effects of a 12-week aquatic dual-task intervention versus conventional aquatic exercise in cognitively preserved older adults accustomed to aquatic environments. Eighty-four participants aged ≥65 years were recruited from the community and screened based on predefined eligibility criteria.

Dual-Task Aquatic Group (GDTA; n = 42): Participants performed motor exercises combined with progressively complex cognitive tasks (e.g., verbal fluency, attention, memory tasks), structured into three progressive phases across 12 weeks.

Conventional Aquatic Exercise Group (GEAC; n = 42): Participants completed a matched program of aquatic motor exercises without cognitive demands.

Both groups received two supervised 45-minute sessions per week in a therapeutic pool. Cognitive and motor functions were assessed immediately before and after the intervention using the Montreal Cognitive Assessment, Mini-Mental State Examination, Timed Up and Go Test, and Berg Balance Scale.

Non-parametric statistical analyses (Wilcoxon and Mann-Whitney tests) were conducted with a significance level of 5%. The GDTA demonstrated significant improvements in cognitive performance, balance, and functional mobility. The GEAC showed significant motor improvements but no cognitive gains. Between-group comparisons confirmed superior cognitive improvement in the GDTA, while motor outcomes did not differ significantly between groups. Adherence to both interventions exceeded 95%.

This study supports the integration of cognitive tasks into aquatic physiotherapy programs for older adults as a strategy to enhance cognitive outcomes while maintaining motor benefits.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 years or older.
* Cognitively preserved, defined as a Mini-Mental State Examination (MMSE) score equal to or above reference values adjusted for education: illiterate ≥16; 1-11 years of schooling ≥23; more than 11 years ≥28.
* Prior experience of 3-6 months with regular aquatic physical therapy (2 sessions per week) to ensure familiarity and adaptation to the aquatic environment.
* Medically cleared to perform moderate-intensity aquatic exercise, confirmed by:
* Orthopedic Assessment: No severe musculoskeletal conditions preventing safe participation.
* Clinical Risk Classification: Low to moderate risk according to the American College of Sports Medicine (ACSM) Risk Stratification.
* Functional Capacity: Duke Activity Status Index score ≥7.

Exclusion Criteria:

* Requirement for walking aids, as this interferes with safety and exercise execution.
* Previous diagnosis of progressive and severe neurological diseases, such as Parkinson's disease, Amyotrophic Lateral Sclerosis, or dementias, that could compromise response to intervention.
* Clinical conditions preventing safe aquatic exercise, including unstable cardiovascular disease, urinary or fecal incontinence, transmissible infectious or dermatological diseases, severe psychiatric disorders, severe respiratory conditions, or acute musculoskeletal limitations.
* Participation in other physical or cognitive training programs during the intervention period.
* Inability to understand or sign the informed consent form.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 84 (Actual)
Dates: Start 2025-04-21 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-10-26 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination | Baseline (pre-intervention) and 12 weeks (post-intervention).
  The Mini-Mental State Examination (MMSE) assesses global cognitive status, including orientation, attention and calculation, memory, language, and visuospatial abilities. The total score ranges from 0 to 30. Education-adjusted cut-offs commonly used to indicate preserved cognition are:
  * Illiterate: ≥16
  * 1-11 years of education: ≥23
  * More than 11 years of education: ≥28
Timed Up and Go Test | Baseline (pre-intervention) and 12 weeks (post-intervention).
  The Timed Up and Go Test evaluates functional mobility, including strength, balance, and gait. The participant stands up from a chair, walks 3 meters, turns, returns to the chair, and sits down. Performance is measured in seconds. Times under 10 seconds generally reflect good mobility, while times above 13.5 seconds indicate increased fall risk.
Montreal Cognitive Assessment | Baseline (pre-intervention) and 12 weeks (post-intervention).
  The Montreal Cognitive Assessment (MoCA) evaluates executive functions, memory, attention, language, visuospatial abilities, abstraction, and orientation. The total score ranges from 0 to 30, with scores below 26 suggesting possible cognitive impairment. One additional point is added for individuals with fewer than 12 years of education.
Berg Balance Scale | Baseline (pre-intervention) and 12 weeks (post-intervention).
  The Berg Balance Scale assesses static and dynamic balance through 14 functional tasks such as standing, reaching, turning, and transferring. Each item is scored from 0 to 4, with a maximum total score of 56. Scores of 40 or below indicate an increased risk of falls.

SECONDARY OUTCOMES:
Adherence to Intervention | Throughout the 12-week intervention.
  Adherence will be calculated based on attendance records of the intervention sessions, expressed as the percentage of completed sessions

CONTACTS AND LOCATIONS:
Overall Officials: Helena S Morgado, BSc, Principal Investigator — Instituto Politécnico de Leiria
Locations (1):
- Clínica de Fisioterapia e Desporto de Pombal, Pombal, Portugal